CLINICAL TRIAL: NCT01904539
Title: An Open-Label, Single-Dose Trial to Assess the Effects of Hepatic Impairment on the Pharmacokinetics of Obeticholic Acid (OCA)
Brief Title: Hepatic Impairment Trial of Obeticholic Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 747-103
Record Dates: First submitted 2013-05-23; First posted 2013-07-22 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — obeticholic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy Volunteer (Experimental): Healthy volunteers receiving a single dose of obeticholic acid 10 mg.
  Interventions: Drug: obeticholic acid 10 mg
- Mild Hepatic Impairment (Experimental): Subjects with mild hepatic impairment defined as Child-Pugh class A receiving a single dose of obeticholic acid 10mg.
  Interventions: Drug: obeticholic acid 10 mg
- Moderate Hepatic Impairment (Experimental): Subjects with moderate hepatic impairment defined as Child-Pugh class B receiving obeticholic acid 10mg.
  Interventions: Drug: obeticholic acid 10 mg
- Severe Hepatic Impairment (Experimental): Subjects with severe hepatic impairment defined as Child-Pugh class C receiving obeticholic acid 10 mg.
  Interventions: Drug: obeticholic acid 10 mg

INTERVENTIONS:
Drug: obeticholic acid 10 mg — Single dose OCA 10mg in each arm
  Other Names: INT-747; 6α-ethyl chenodeoxycholic acid; 6-ECDCA

SUMMARY:
This is a phase 1 study to evaluate the safety of a single 10 mg dose of obeticholic acid (OCA) in healthy volunteers and patients with liver disease.

ELIGIBILITY:
Subject Inclusion Criteria All Subjects

* Female and male subjects ≥ 18 years of age
* Subjects will have a minimum body weight of 45 kg or body mass index (BMI)> 18 kg/m2.
* Contraception: Female subjects must be postmenopausal, surgically sterile, or if premenopausal, be prepared to use ≥ 1 effective method of contraception during the trial and until at least 30 days after administration of OCA.
* Subjects must provide written informed consent and agree to comply with the trial protocol.

Subjects with Hepatic Impairment:

* Evidence of hepatic disease

  1. Score ≥ 2 on one of the Child-Pugh parameters, or
  2. Histological diagnosis of cirrhosis or presence of esophageal varices, or
  3. Abnormal alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) levels
* Subjects will satisfy the criteria of the modified Child-Pugh classification for hepatic impairment during Screening:

  1. Mild hepatic impairment: Class A (Child-Pugh Scores 5-6 points)
  2. Moderate hepatic impairment: Class B (Child-Pugh Scores 7-9 points)
  3. Severe hepatic impairment: Class C (Child Pugh Scores 10-15 points)

Healthy volunteers:

* Absence of clinically-relevant abnormalities identified by a detailed medical history, full physical examination, 12-lead ECG
* Clinical laboratory tests within the normal reference range
* Subjects must be within ± 10 years of the mean age and within 20% of the mean BMI of the hepatic impaired subjects (Child-Pugh category A, B, and C)

Subject Exclusion Criteria All Subjects

* Positive test for human immunodeficiency virus (HIV)-1 or HIV-2 at screening
* Presence or history of malignancy, with the exception of basal cell carcinoma
* Received an investigational drug, including OCA, within 30 days or t½=5 prior to dosing
* Blood or plasma donation within 30 days prior to dosing
* History of non-compliance to medical regimens, or subjects who are considered to be potentially unreliable
* Presence or history of clinically significant cardiac arrhythmias that may prohibit the subject from participating in the trial
* Female subjects who are pregnant or lactating
* Subjects who have irritable bowel disease or other GI disorders that have the potential to alter drug or bile acid absorption.
* Subjects who have a history of gall bladder removal, gastric bypass or other GI surgery that may affect drug absorption or the enterohepatic circulation.

Subjects with Hepatic Impairment

* History of alcohol or drug abuse 3 months prior to dosing
* In the opinion of the Investigator and medical monitor, fluctuating or rapidly deteriorating hepatic function within the screening period
* In the opinion of the Investigator, any evidence of additional severe or uncontrolled systemic disease or evidence of any other significant clinical disorder or laboratory finding likely to affect the conduct of the trial or interpretation of the data
* Subjects who have a transjugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting
* Subjects with Wilson's disease, alpha-1 antitrypsin deficiency, glycogen storage diseases and galactosemia
* Heavy smoker or use of tobacco or nicotine products

Healthy Volunteers

* Presence of significant uncontrolled disease that will complicate execution of the trial or interfere with the absorption, distribution, metabolism, or excretion of drugs via the gut
* Evidence of chronic or acute liver disease as documented by medical history, physical examination or diagnostic tests that it likely to affect the conduct of the trial or interpretation of the data
* History of and/or current alcohol abuse (defined as consumption of more than 210 mL of alcohol per week; or the equivalent of fourteen 4-oz glasses of wine, or fourteen 12-oz cans/bottles of beer or wine coolers per week) or drug abuse within the prior two years
* Smoke or use tobacco or nicotine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of OCA and conjugates | Up to 48 hours
  maximum concentration
Area under the concentration versus time curve from time 0 to the last sampling time with measurable analyte concentration (AUCt) of OCA and conjugates | Post-dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, and 216 hours post-dose
Time to Cmax (Tmax) of OCA and conjugates | Up to 48 hours
Area under the concentration versus time curve from time 0-24 hours with measurable analyte concentration of OCA and conjugates. (AUC 0-24) | 24 hours

SECONDARY OUTCOMES:
Urine concentration of unchanged OCA and conjugates | 0, 6, 12, 24, 30 hours
Amount of OCA and conjugates excretion in urine | -6to 0, 0 to 6, 6 to 12, 12 to 24, and 24 to 30 hours
Total amount of OCA and conjugates excreted in urine | 0 to 30 hours
Protein Binding | 0, 0.75, 1.5, 6, and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Shapiro, MD, Study Director — Intercept Pharmaceuticals
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

REFERENCES:
- [Derived] Edwards JE, LaCerte C, Peyret T, Gosselin NH, Marier JF, Hofmann AF, Shapiro D. Modeling and Experimental Studies of Obeticholic Acid Exposure and the Impact of Cirrhosis Stage. Clin Transl Sci. 2016 Dec;9(6):328-336. doi: 10.1111/cts.12421. Epub 2016 Oct 15. PMID 27743502